CLINICAL TRIAL: NCT06275919
Title: Regorafenib for Recurrent Grade 2 and 3 Meningioma. A Multicenter, Randomized Phase II Study (MIRAGE Trial)
Brief Title: Regorafenib for Recurrent Grade 2 and 3 Meningioma (MIRAGE Trial)
Acronym: MIRAGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-BT-1-2023 MIRAGE
Record Dates: First submitted 2024-02-07; First posted 2024-02-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Meningioma, Malignant
MeSH Terms: conditions — Meningioma | interventions — regorafenib; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (interventional arm) (Experimental): REGORAFENIB 40 mg tablets once daily (160 mg/die), 3 weeks on, 1 week off, until disease progression or unacceptable toxicity
  Interventions: Drug: Regorafenib 40 MG Oral Tablet
- Arm B (control arm) (Active Comparator): Local Standard of Care until disease progression or unacceptable toxicity
  Interventions: Drug: Local Standard of Care

INTERVENTIONS:
Drug: Regorafenib 40 MG Oral Tablet — REGORAFENIB 40 mg tablets once daily (160 mg/die), 3 weeks on, 1 week off, until disease progression or unacceptable toxicity
  Arms: Arm A (interventional arm)
Drug: Local Standard of Care — In this setting there are not drugs with indication. Every site will treat patients as per their experience.
  Arms: Arm B (control arm)

SUMMARY:
The focus of this study will be to investigate whether Regorafenib demonstrates antitumor activity against recurrent grade II or III meningiomas.

Small trials and case series suggest clinical relevant activity of several VEGF inhibitors such as sunitinib, bevacizumab and valatinib reporting a 6m-PFS rate of 42-64%. Indeed, VEGF and VEGF receptors (VEGFR) are regularly overexpressed in meningiomas and can correlate with outcome.

Regorafenib inhibits angiogenic receptor tyrosine kinases (RTKs) and is highly selective for VEGFR1/2/3; moreover Regorafenib inhibits PDGFRB, FGFR1 and oncogenic intracellular signalling cascades involving c-RAF/RAF1 and BRAF highly expressed in meningiomas.

Noteworthy, Regorafenib showed antitumor activity in vitro and in vivo in a recent study; indeed, Regorafenib showed significant inhibition of meningioma cell motility and invasion and in vivo, mice with orthotopic meningioma xenografts showed a reduced volume of signal enhancement in MRI following Regorafenib therapy; this translated in a significantly increased overall survival time (p<0.05) for Regorafenib treated mice.

Moreover, Regorafenib showed good efficacy in different cancer types, such as colorectal cancer, GIST, hepatocellular carcinoma and glioblastoma (REGOMA trial) , maintainingmaintaining a good quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
* Patients capable of taking oral medication
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
* Histological diagnosis of grade 2 or grade 3 meningioma according to the WHO 2021 classification
* Radiologically documented progression of any existing tumor with an estimated planar growth >25% (bidirectional) in the last 12 months or appearance of new lesions
* Ineligible for further surgery and/or radiotherapy
* at least 1 Measurable lesion (minimum 10 x 10mm) on baseline MRI
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 to 1 (or KPS ³70)
* Male or female ≥ 18 years of age
* Subjects must have life expectancy of at least 6 months
* Paraffin-embedded tumor tissue available (mandatory)
* Dosage of dexamethasone or equivalent steroid within 7 days prior the randomization ≤4mg/die
* Stable or decreasing dosage of steroids for 7 days prior to the randomization.
* Adequate cardiac function and adequate liver, renal and hematological function
* Subject must have the following laboratory values at screening within 14 days before starting Regorafenib:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if subject received pegfilgrastim).
* Hemoglobin (Hgb) ≥10 g/dL
* Platelet count (plt) ≥100x 109/L
* Serum potassium concentration within normal range, or correctable with supplements
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamate pyruvic transaminase (SGPT)/alanine aminotransferase (ALT) ≤ 3.0 x Upper Limit of Normal (ULN).
* Serum total bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN or measured glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m2 using an exogenous filtration marker such as iohexol, inulin, 51Cr EDTA or 1125 iothalamate, or creatinine clearance of ≥ 50 mL/min using Cockroft-Gault equation.
* Serum albumin > 3.5 g/dL
* PT (or INR) and APTT within normal range
* For women who are not postmenopausal (i.e., < 2 years after last menstruation) or surgically sterile (absence of ovaries and/or uterus) and who are sexually active: agreement to use an adequate method of contraception (oral contraceptives, intrauterine contraceptive device, or barrier method of contraception in conjunction with spermicidal jelly) during the Treatment period and for at least 6 months after the last dose of study drug.
* For male patients who are partners of premenopausal women: agreement to use a barrier method of contraception during the Treatment period and for at least 6 months after the last dose of study drug.
* Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to participate.
* 19. Patients with measurable, progressive meningioma who received radiation therapy are potentially eligible but need to show evidence of progression at least 24 weeks from completion of radiation therapy.

Exclusion Criteria:

* Prior antineoplastic therapy for meningioma
* Subject incapacitated to understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted
* Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort)
* Are taking strong UGT1A9 inhibitors (e.g. mefenamic acid, diflunisal and niflumic acid)
* Receiving additional, concurrent, active therapy for Meningioma outside of the trial.
* Disease outside the brain (ie. spinal cord or bone or metastasis to a distant organ)
* Candidate for urgent palliative intervention for primary disease (e.g., impending herniation) as judged by the Investigator
* History of allergy or hypersensitivity to any of the study treatments or any of their excipients.
* In the presence of therapeutic intent to anticoagulate the patient:,INR or PT and aPTT not within therapeutic limits (according to the medical standard in the institution)
* Unable or unwilling to undergo brain MRI scans with intravenous (IV) gadolinium
* History of another malignancy in the previous 3 years, with a disease-free interval of< 3 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
* Serious, non-healing wound, ulcer, bone fracture, or abscess.
* Any cerebrovascular accident (including transient ischemic attacks) within the last 6 months prior to initiation of study treatment.
* Have an ongoing infection with severity of Grade 2 or above (CTCAE 5.0)
* Any hemorrhage or bleeding event that is ≥ Grade 3 based on the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE), Grade 2 intracranial hemorrhage, or persistent thrombotic/embolic event within 4 weeks prior to the start of study medication.
* Uncontrolled or severe cardiac disease (e.g., history of unstable angina, myocardial infarction, coronary stenting, or bypass surgery within the last 6 months prior to initiation of study treatment), symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia (including atrial flutter/fibrillation), requirement for inotropic support or use of devices for cardiac conditions (e.g.,pacemakers/defibrillators), or hypertension (participants with systolic blood pressure[BP] of > 160 mmHg or diastolic BP of > 100 mmHg despite optimal medical management are to be excluded).
* History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis, or symptomatic pleural effusion.
* Active, known, or suspected auto-immune disease, including systemic lupus erythematosus, Hashimotos thyroiditis, scleroderma, polyarteritis nodosa, or auto-immune hepatitis.
* Known history of hepatitis B, human immunodeficiency virus (HIV), or active hepatitis C infection requiring treatment with antiviral therapy. Note: HIV testing is not required in the absence of clinical suspicion.
* History of bleeding diathesis (irrespective of severity).
* Uncontrolled intercurrent illness including (e.g., symptomatic ascites), but not limited to ongoing or active infection.
* Persistent ≥ Grade 3 Lipase (> 2.0 - 5.0 x upper limit of normal [ULN] with signs or symptoms; > 5.0 x ULN and asymptomatic).
* Persistent proteinuria > 3.5 g/24 hours measured by urine protein creatinine ratio from a random urine sample (≥ Grade 3, CTCAE 5.0)
* Have any malabsorbition condition
* Any condition that could make the subject noncompliant with the study procedures and/or study requirements, as judged by the Investigator (for example: cognitive impairment, psychiatric illness, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 36 months
  The progression free survival (PFS) will be determined as the time from the date of enrolment to the date of disease progression determined using RANO criteria or to the date of death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 30 months
  The overall survival (OS) will be determined as the time from the date of enrolment to the date of death from any cause.
Objective response rate (ORR) | Up to 30 months
  The objective response rate (ORR) will be defined as the percentage of patients with complete response (CR) and partial response (PR) determined using modified Macdonald criteria.
Patient Reported Outcomes (PROs) | Up to 30 months
  Quality of life will be assessed by EORTC QLQ-C30 questionnaire.
Patient Reported Outcomes (PROs) | Up to 30 months
  Quality of life will be assessed by the QLQBN20 questionnaire.
Toxicity during treatment | Up to 30 months
  Toxicity during the treatment will be recorded and graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v.5.
Disease control rate (DCR) | Up to 30 months
  The disease control rate (DCR) will be defined as the percentage of patients with complete response (CR), partial response (PR) and stable disease (SD) determined using modified Macdonald criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lombardi, MD, Principal Investigator — Istituto Oncologico Veneto IOV IRCCS
Locations (16):
- Italy (16):
  - IRST Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola, Forlì-Cesena
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina, Italia/Messina
  - Humanitas Cancer Center, Rozzano, Milano
  - Ospedale San Paolo, Bari
  - Ospedale Bellaria - AUSL Bologna, Bologna
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Policlinico San Martino, Genova
  - Spedali Riuniti, Livorno
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale del Mare, Napoli
  - Istituto Oncologico Veneto, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - IRCCS Istituto Tumori Regina Elena, Roma
  - Policlinico Umberto I - Università Sapienza Roma, Roma
  - A.O.U. Città della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bosio A, Cerretti G, Padovan M, Del Bianco P, Polano M, Mandruzzato S, Indraccolo S, Manara R, Librizzi G, Caccese M, Corra M, Maccari M, Lonardi S, De Salvo GL, Lombardi G. Regorafenib versus local standard of care in patients with grade 2-3 meningioma no longer eligible for loco-regional treatments: a phase II randomized controlled trial (the MIRAGE study). Trials. 2025 Aug 4;26(1):268. doi: 10.1186/s13063-025-08997-2. PMID 40759981